CLINICAL TRIAL: NCT06889168
Title: A Phase 1, Randomized, Double-blinded, Placebo Controlled, Trial Evaluating the Long-term Safety and Tolerability of Imatinib for the Treatment of Lymphangioleiomyomatosis [LAMP-2 Trial]
Brief Title: Evaluating the Long-term Safety and Tolerability of Imatinib in Patients With Lymphangioleiomyomatosis (LAM)
Acronym: LAMP-2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jeanine D'Armiento, Professor of Medicine in Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAT1955
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lymphangioleiomyomatosis (LAM); Lymphangioleiomyomatosis
Keywords: LAM; LAMP-2; Imatinib
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imatinib Mesylate Group (Active Comparator): This group will receive imatinib mesylate over the course of the trial.
  Interventions: Drug: Imatimib Mesylate
- Placebo Group (Placebo Comparator): This group will receive placebo over the course of the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imatimib Mesylate — Participants will take Imatinib mesylate (imatinib), an FDA approved drug for leukemia, orally 400 mg (twice daily)
  Other Names: Gleevec®; imatinib
  Arms: Imatinib Mesylate Group
Drug: Placebo — Placebo will be administered in the same dosage and manner as the study drug. The placebo looks like the study drug but contains no active ingredients.
  Arms: Placebo Group

SUMMARY:
Lymphangioleiomyomatosis (LAM) is a rare cystic lung disease that appears to behave like a slowly growing cancer. Since clinical progression is very slow, new blood tests have been used to speed the time required to find safe and effective medications. A large National Institute of Health study called MILES showed that sirolimus (also known as Rapamycin) improved lung function in individuals with LAM. Since most individuals with LAM and impaired lung function are now on sirolimus, future studies may prove more difficult. Laboratory studies suggested that Imatinib mesylate (imatinib), an FDA-approved drug for leukemia, initiates LAM cell death. A pilot trial with imatinib titled "Imatinib Mesylate for the treatment of Lymphangioleiomyomatosis" - (LAMP-1) was funded by the Department of Defense in 2016, and documented (1) the safety of use of tyrosine kinase inhibitors in patients with LAM; (2) the safety of concurrent use of tyrosine kinase and mTOR inhibitors; and, (3) short term variability in vascular endothelial growth factor D (VEGF-D) - a LAM biomarker, as a response to therapies. Due to the short-term LAMP-1 trial, LAMP-2 will be a longer-term 6-month clinical study evaluating the safety and tolerability of imatinib in patients with LAM. Patients that participate in the trial will come in for 5 office visits and check-up phone calls every 2 weeks over the course of 6 months.

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis (LAM) is a rare cystic lung disease that is due to a very slow growing cancer that proliferates via unopposed activity of the mTOR pathway. A large NIH study (MILES) found that sirolimus (Rapamycin) that inhibits the mTOR pathway improved lung function and quality of life compared to placebo in LAM. Sirolimus has been shown to cause growth suppression but not apoptosis of LAM cells in culture. Additionally, not all patients with LAM have a clinical effect with sirolimus. Recently, imatinib mesylate has been shown to induce LAM cell apoptosis, raising the possibility of more lasting therapy for LAM. Currently, most LAM patients are on sirolimus and attempts to find sirolimus naive patients have not been successful for other studies. LAM cells use the mesenchymal PDGF receptor pathway for proliferation, similar to certain leukemias and slow growing neoplasms. Laboratory studies suggested that Imatinib mesylate (imatinib), an FDA approved drug for leukemia, initiates LAM cell death. A pilot trial with imatinib (LAMP-1) was funded by the DOD in 2016, and documented (1) the safety of use of tyrosine kinase inhibitors in patients with LAM; (2) the safety of concurrent use of tyrosine kinase and mTOR inhibitors; and, (3) short term variability in VEGF-D as a response to therapies. Concurrent cell-based research studies during this time showed equally efficacious tumoricidal activity of nilotinib in vitro. Due to the short-term LAMP-1 trial, the investigators propose a longer-term clinical study evaluating the safety and tolerability of imatinib in patients with LAM.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 through 64 years of age (inclusive)
* Pulmonary Function Test (PFT) with following criteria:

  1. DLCO >20% predicted and FVC <90% OR
  2. Post bronchodilator FEV1 between 30% and 90% predicted.
* Confirmed or possible diagnosis of LAM
* Willing to avoid grapefruit juice and St. John's wort while in the study
* Able and willing to comply with the study procedures

Exclusion Criteria:

* Women who have or will undergo a transplant
* Women who will undergo surgery
* Women who are currently pregnant or plan on a pregnancy
* Women who are currently breast feeding or lactating
* Dementia or other cognitive dysfunction that, in the opinion of the investigator, would prevent the participant from consenting to the study or completing study procedures
* Currently taking any of the following medications:

  * Antifungal Medications: Ketoconazole; Itraconazole ; Voriconazole.
  * Antibiotics for bacterial infections: Clarithromycin.
  * Analgesics to treat headaches/migraines: Dihydroergotamine; Dihydroergotamine intranasal
  * Antiretroviral protease inhibitors used in human immunodeficiency virus (HIV) infections: Atazanavir ; Nelfinavir; Indinavir; Ritonavir; Saquinavir
  * Anti-epileptic or seizure medications: Carbamazepine, Fosphenytoin; Oxcarbamazepine; Phenobarbital ; Phenytoin; Primidone
  * Anti-depressant medications: Nefazodone; St. John's wort
  * Targeted cancer drugs: Regorafenib; Venetoclax ; Cobimetinib
  * Ivabradine (used to treat chronic heart failure); Telithromycin (used to treat community acquired pneumonia); Lomitapide (treatment of familial hypercholesterolemia); Lonafarnib (Hutchinson-Gilford progeria syndrome); conivaptan (treat low sodium levels); flibanserin (management of hypoactive sexual desire disorder (HSDD)); Naloxegol (opioid-induced constipation); Warfarin (prevent blood clots); Lurasidone (schizophrenia and bipolar depression); Eliglustat (treatment of Gaucher's disease).
* Non English speaking, illiterate, or other vulnerable persons will not be included among study subjects.
* Any condition that in the opinion of the investigator might adversely influence the study outcome.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 1 year
  To observe and compare the occurrence of adverse events experienced by participants receiving imatinib mesylate compared to placebo throughout the duration of the study.

SECONDARY OUTCOMES:
Change in VEGF-D between study groups | Baseline, 6 months
  To compare the change in the log-transformed level of VEGF-D from baseline to 6 months between imatinib mesylate and placebo groups.
Change in Forced Vital Capacity (FVC) between study groups | Baseline, 6 months
  To compare the change in Forced Vital Capacity (FVC) from baseline to 6 months between imatinib mesylate and placebo groups.
Change in percent Forced Expiratory Volume in One Second (FEV1) between study groups | Baseline, 6 months
  To compare the change in the percent predicted FEV1 (Forced expiratory volume in one second) using "GLI other" standards from baseline to 6 months between imatinib mesylate and placebo groups.
Change in St. George Respiratory Questionnaire (SGRQ) score between study groups | Baseline, 6 months
  To compare the change in the total score of the St. George Respiratory Questionnaire (SGRQ) from baseline to 6 months between imatinib mesylate and placebo groups. Scores range from 0 to 100, with 0 representing no health impairment and 100 representing maximum health impairment.

OTHER OUTCOMES:
Change in High Mobility Group AT-Hook2 (HMGA2) between study groups | 1 year
  To compare the change in expression of the neural crest biomarker HMGA2 (High Mobility Group AT-Hook2) between imatinib and placebo groups in the entire group, and in those not on sirolimus.
Change in percent Forced Expiratory Volume in One Second (FEV1) | 1 year
  To compare the change in the percent predicted FEV1 between imatinib and placebo groups in those not on sirolimus.
Change in Modified Medical Research Council (mMRC) Dyspnea Score | 1 year
  To compare the change in mMRC (Modified Medical Research Council) Dyspnea score between imatinib and placebo groups in the entire group and in those not on sirolimus. The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4. A higher score indicates a higher degree of disability due to breathlessness.
Change in 6 Minute Walk Test (6MWT) | 1 year
  To compare the change in the 6MWT (6 Minute Walk Test) distance between imatinib and placebo groups in the entire group and in those not on sirolimus. The 6MWT measures how far a participant can walk in 6 minutes.
Change in EuroQol 5 Dimension (EQ5D) | 1 year
  To compare the change in EQ5D scores between imatinib and placebo groups in the entire group and in those not on sirolimus. The EQ-5D (EuroQol 5 Dimension) is a questionnaire designed to measure a person's health-related quality of life by assessing their self-reported experiences across five key dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scoring is based on a scale of 0-100, 0 being the worst imaginable health state and 100 being the best imaginable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine D'Armiento, MD, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina